CLINICAL TRIAL: NCT02901457
Title: "The Healthy Body Image" (HBI) Program: A Program to Promote a Positive Body Image. A School-based Randomized Controlled Trial
Brief Title: "The Healthy Body Image" (HBI) Program: A Program to Promote a Positive Body Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other); Norwegian Extra Foundation for Health and Rehabilitation (Other); University of Tromso (Other); University College of Southeast Norway (Other); University of Agder (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JCSB
Record Dates: First submitted 2016-04-24; First posted 2016-09-15 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2021-08

CONDITIONS: Quality of Life; Eating Behaviors; Physical Activity
Keywords: Body Image
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Body Image (Experimental): Students receive the Healthy Body Image intervention containing 3x90 minutes of interactive workshops with the addition of related homework after each workshop.
  Interventions: Other: The "Healthy Body Image" intervention
- Control group (No Intervention): Students do not receive the intervention program.

INTERVENTIONS:
Other: The "Healthy Body Image" intervention — Interactive workshops (3 x 90 minutes) include training techniques to increase media literacy, enhance self-esteem, positive body image, awareness of perfectionism, and include discussions related to truths and myths related to life style factors. Homework is an extension of each workshop that is simple and not time-consuming tasks to increase reflection and awareness of how all the mentioned factors are a part of their lives.
  Other Names: Healthy Body Image
  Arms: Healthy Body Image

SUMMARY:
Too many Norwegian adolescents experience severe body dissatisfaction (40-70 %), and strive to accomplish the "perfect body". At the same time, only 50 % meet the government's recommendations on physical activity and intake of fruits and vegetables. Also, 14-24 % has unhealthy sleeping habits. Optimizing these lifestyle factors is associated with physical and psychological health. These factors, along with the pressure to obtain the "perfect" body, are threatening the adolescent's physical and psychological health, jfr. Meld St nr 19. It is now a need for knowledge on how the investigators can contribute to promote positive body experience among the adolescents.

It has recently, through a controlled study on elite youth athletes at Norwegian sports high schools, been shown that it is possible to change eating habits, improve body image and reduce new cases of eating disorder. It is now desirable to test an adapted program through a school-based program at regular Norwegian high school students (12th grade). Today, no controlled, school-based intervention studies with long-term follow-up have been conducted.

The main aim of this project is to investigate if it is possible, through a school-based intervention program (Healthy Body Intervention), to promote positive body image, increase physical activity level, and healthy eating and sleeping habits in both boys and girls at Norwegian high schools.

The intervention program will contribute with new evidence-based knowledge on the effect of an adapted health-promoting program.

DETAILED DESCRIPTION:
The design is a school-based randomized controlled trial (RCT) intervention, using the methods questionnaire and interview to obtain data. Based on statistical power analyses, all high schools in Oslo and Akershus County will be asked to participate in the study. After the schools have responded, consenting schools will be stratified (by size and geographical affiliation) and randomized to the intervention or the control condition. To minimize contamination biases within schools, the investigators prepare a cluster-randomized design.The population should contain 17-20 schools (1400 students at 2nd year). Data collection is conducted through pre-test and post-test 1, 2, and 3 (acute, 3, and 12 month post-intervention). At post-test 1, a selection is invited to participate in an interview about feasibility in addition to the questionnaire. It is an intervention for students containing interactive lecturers with discussion, team work, discussions and home assignments.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian high schools
* High schools located in either Oslo or Akershus County
* Students in the 2nd grade fall 2016
* Students within academic specialization education programs
* Teachers teaching included students in Norwegian, Social studies, Physical education, and contact teachers
* School nurses working at the randomly selected schools
* School administrators at randomly selected schools

Exclusion Criteria:

* Schools that follow foreign school systems
* Students within vocational education programs
* School departments connected to prison

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4193 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Proximal and distal effect of the "Healthy Body Intervention" (HBI) program on change in positive body image | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  Participants are asked to respond to questions by choosing from different responses presented on a likert scale. Positive body image is assessed by the Experience of Embodiment Scale.

SECONDARY OUTCOMES:
Proximal and distal effect of the HBI program on change in self-esteem | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  Participants are asked to respond to questions by choosing from different responses presented on a likert scale. The scale used is the Rosenberg Self-esteem scale.
Proximal and distal effect of the "Healthy Body Intervention" (HBI) program on change in the prevalence of students meeting the recommendations for health promoting physical activity. | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  The outcome will be measured through a self-developed Physical Activity level/habit questionnaire, including choosing a specific response on a likert scale and response through open ended questions.
Experience of the intervention program and the feasibility of running the HBI program in schools. | Post-test is planned within first week after intervention
  To measure the outcome, a self-developed interview guide in addition to a self-developed questionnaire asking students and school staff about the experience of the intervention program and the feasibility of the intervention. When answering the questionnaire, participants are asked to respond by choosing a response on a likert scale.
Proximal and distal effect of the HBI program on change in eating behavior (nutrition intake | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  The outcome will be measured through a self-developed Food frequency questionnaire where responses are chosen from a likert scale.
Proximal and distal effect of the HBI program on change in sleeping quality and sleep patterns | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  The outcome is measured through The Bergen Insomnia Scale, 6 items and 3 items assessing delayed sleep phase and by asking the participants (using a likert scale) how many hours of sleep they usually get per night during a normal weekday and a weekend day.
Proximal and distal effect of the HBI program on change in academic achievements | Participants are asked to complete the questions included in the questionnaire package at post-tests planned at week 1, 3 months and 12 months after intervention
  Participants are asked to choose the correct grade they received on their last report card, from a scale presenting the possible grades.
Proximal and distal effect of the "Healthy Body Intervention" (HBI) program on change in health related quality of life | Participants are asked to complete the questionnaire containing all the below presented measures at post-tests planned at week 1, 3 months and 12 months after intervention
  Participants are asked to respond to questions by choosing from different responses presented on a likert scale. Health related quality of life will be assessed through the "Screening for and Promotion of Health Related Quality of Life in Children an Adolescents - a European Public Health Perspective - 10" (KIDSKREEN-10).
Proximal and distal effect of the HBI program on change in symptoms of eating disorders | Participants are asked to complete the questionnaire at post-tests planned at week 1, 3 months and 12 months after intervention
  Symptoms of eating disorders is assessed by the Eating Disorder Examination Questionnaire - 11 (EDE-Q 11)

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, Phd, Study Chair — Norwegain School of Sports Sciences
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strand BH, Dalgard OS, Tambs K, Rognerud M. Measuring the mental health status of the Norwegian population: a comparison of the instruments SCL-25, SCL-10, SCL-5 and MHI-5 (SF-36). Nord J Psychiatry. 2003;57(2):113-8. doi: 10.1080/08039480310000932. PMID 12745773
- [Background] Andersen JR, Natvig GK, Haraldstad K, Skrede T, Aadland E, Resaland GK. Psychometric properties of the Norwegian version of the Kidscreen-27 questionnaire. Health Qual Life Outcomes. 2016 Apr 9;14:58. doi: 10.1186/s12955-016-0460-4. PMID 27062022
- [Background] Rosenberg M. Society and the Adolescent Self-Image. Princeton, NJ: Princeton University Press; 1965.
- [Background] Pallesen S, Hetland J, Sivertsen B, Samdal O, Torsheim T, Nordhus IH. Time trends in sleep-onset difficulties among Norwegian adolescents: 1983--2005. Scand J Public Health. 2008 Nov;36(8):889-95. doi: 10.1177/1403494808095953. PMID 19004908
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Friborg O, Reas DL, Rosenvinge JH, Ro O. Core pathology of eating disorders as measured by the Eating Disorder Examination Questionnaire (EDE-Q): the predictive role of a nested general (g) and primary factors. Int J Methods Psychiatr Res. 2013 Sep;22(3):195-203. doi: 10.1002/mpr.1389. Epub 2013 Aug 19. PMID 24038315
- [Background] Sandoz EK, Wilson, K.G., Merwin, R.M., Kellum, K.K. Assessment of body imageflexibility: The Body Image-Acceptance and Action Questionnaire. Journal of Contextual Behavioral Science. 2013:39-48
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Smolak L, Murnen SK. Drive for leanness: assessment and relationship to gender, gender role and objectification. Body Image. 2008 Sep;5(3):251-60. doi: 10.1016/j.bodyim.2008.03.004. Epub 2008 Jun 26. PMID 18585105
- [Background] Smolak L, & Piran, N. . Gender and the prevention of eating disorders. In: G. McVey MPL, N. Piran & H. B. Ferguson editor. Preventing eating-related and weight-related disorders: Collaborative research, advocacy, and policy change. Waterloo, ON: Wilfred Laurier Press; 2012. p. 201-24.
- [Derived] Sundgot-Borgen C, Friborg O, Kolle E, Torstveit MK, Sundgot-Borgen J, Engen KME, Rosenvinge JH, Pettersen G, Bratland-Sanda S. Does the Healthy Body Image program improve lifestyle habits among high school students? A randomized controlled trial with 12-month follow-up. J Int Med Res. 2020 Mar;48(3):300060519889453. doi: 10.1177/0300060519889453. Epub 2019 Dec 5. PMID 31802697
- [Derived] Sundgot-Borgen C, Bratland-Sanda S, Engen KME, Pettersen G, Friborg O, Torstveit MK, Kolle E, Piran N, Sundgot-Borgen J, Rosenvinge JH. The Norwegian healthy body image programme: study protocol for a randomized controlled school-based intervention to promote positive body image and prevent disordered eating among Norwegian high school students. BMC Psychol. 2018 Mar 6;6(1):8. doi: 10.1186/s40359-018-0221-8. PMID 29510762